CLINICAL TRIAL: NCT02471235
Title: Effect of Short Course Out-patient Pulmonary Rehabilitation on the Activity and Frequency of Exacerbations of Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Short-course Out-patient Pulmonary Rehabilitation and COPD Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012 COPD care program_02
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The physiotherapist will provide every patient an individualized physical training programme that fits their cardiopulmonary status. Patients will have the training as out-patient in the physiotherapy department for 4-8 sessions, 2 hours each time, 1-2 times weekly. Home exercise will be taught. Our case manager will give phone calls to the subject every 2 weeks to provide support and reinforcement for having continuous exercise at home for one year. Patients will be invited to attend reinforcement out-patient physiotherapy training once very month or every 2 months if they are willing to attend.
  Interventions: Behavioral: Physiotherapy
- Control group (No Intervention): The control group will receive no physiotherapy training by physiotherapist and no phone calls from case manager for reinforcement of home exercise. .

INTERVENTIONS:
Behavioral: Physiotherapy — Pulmonary rehabilitation
  Arms: Intervention group

SUMMARY:
This study assessed whether a short course pulmonary rehabilitation programme with periodic reinforcement exercise training and phone call reminders would help to increase physical activity in COPD patients and also decrease readmissions for AECOPD.

DETAILED DESCRIPTION:
Objectives: Chronic obstructive pulmonary disease (COPD) is a disease with significant morbidity and incurs heavy utilization of healthcare resources. The direct cost of hospital admissions related to COPD is the single largest source of expenditure in the public hospital system. This study assessed whether a short course pulmonary rehabilitation programme with periodic reinforcement exercise training and phone call reminders would help to increase physical activity in COPD patients and also decrease readmissions for AECOPD.

Hypothesis: The above programme can reduce readmissions for AECOPD

Design: Randomised control trial. Patients will be randomised to the intervention or usual care group

Subjects: Patients discharged from hospital after an episode of acute exacerbation of COPD

Study instruments: Activity monitor, quality of life questionnaire

Interventions: The Intervention group will receive a short course pulmonary rehabilitation training as out-patient in the physiotherapy department for 4-8 sessions, 2 hours each time, 1-2 times weekly. The training is scheduled in the way that each subject would have at least 4-8 weeks supervised training by trained physiotherapist. Home exercise will be taught and the case manager will give phone calls to the subject every 2 weeks to provide support and reinforcement for having continuous exercise at home for one year. Patients will be invited to attend reinforcement out-patient physiotherapy training once very month or every 2 months if they are willing to attend.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD exacerbations

Exclusion Criteria:

1. History of asthma, lung resection or other significant pulmonary disease like pulmonary fibrosis.
2. Active infection like pulmonary tuberculosis
3. Unable to complete assessment due to physical and/or cognitive impairment
4. Completed a pulmonary rehabilitation program in the previous 24 months.
5. Having short life expectancy like subjects with terminal malignancy or intractable heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
hospital readmissions | 12 months
  The primary endpoint is the hospital readmissions

SECONDARY OUTCOMES:
Activity measure by the activity monitor | 12 months
mortality | 12 months
lung function | 12 months
Body mass index | 12 months
exercise capacities | 12 month
  by 6 minute walk test
Quality of life questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fanny WS Ko, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, N.T.
  - Prince of Wales Hospital, Shatin

REFERENCES:
- [Background] Global initiative for chronic obstructive lung disease. Global strategy for the diagnosis, management and prevention of chronic obstructive pulmonary disease. 2013 http://www.goldcopd.org/uploads/users/files/GOLD_Report_2013_Feb20.pdf Access date: 28 Oct 2013.
- [Background] Buist AS, McBurnie MA, Vollmer WM, Gillespie S, Burney P, Mannino DM, Menezes AM, Sullivan SD, Lee TA, Weiss KB, Jensen RL, Marks GB, Gulsvik A, Nizankowska-Mogilnicka E; BOLD Collaborative Research Group. International variation in the prevalence of COPD (the BOLD Study): a population-based prevalence study. Lancet. 2007 Sep 1;370(9589):741-50. doi: 10.1016/S0140-6736(07)61377-4. PMID 17765523
- [Background] Ko FW, Hui DS, Lai CK. Worldwide burden of COPD in high- and low-income countries. Part III. Asia-Pacific studies. Int J Tuberc Lung Dis. 2008 Jul;12(7):713-7. PMID 18544193
- [Background] Chan-Yeung M, Lai CK, Chan KS, Cheung AH, Yao TJ, Ho AS, Ko FW, Yam LY, Wong PC, Tsang KW, Lam WK, Ho JC, Chu CM, Yu WC, Chan HS, Ip MS, Hui DS, Tam CY; Hong Kong Thoracic Society. The burden of lung disease in Hong Kong: a report from the Hong Kong Thoracic Society. Respirology. 2008 Nov;13 Suppl 4:S133-65. doi: 10.1111/j.1440-1843.2008.01394.x. PMID 18945323
- [Background] Ko FW, Woo J, Tam W, Lai CK, Ngai J, Kwok T, Hui DS. Prevalence and risk factors of airflow obstruction in an elderly Chinese population. Eur Respir J. 2008 Dec;32(6):1472-8. doi: 10.1183/09031936.00058708. Epub 2008 Aug 6. PMID 18684847
- [Background] Ko FW, Ip M, Chan PK, Fok JP, Chan MC, Ngai JC, Chan DP, Hui DS. A 1-year prospective study of the infectious etiology in patients hospitalized with acute exacerbations of COPD. Chest. 2007 Jan;131(1):44-52. doi: 10.1378/chest.06-1355. PMID 17218555
- [Background] Ko FW, Ip M, Chan PK, Chan MC, To KW, Ng SS, Chau SS, Tang JW, Hui DS. Viral etiology of acute exacerbations of COPD in Hong Kong. Chest. 2007 Sep;132(3):900-8. doi: 10.1378/chest.07-0530. Epub 2007 Jun 15. PMID 17573516
- [Background] Ko FW, Tam W, Wong TW, Chan DP, Tung AH, Lai CK, Hui DS. Temporal relationship between air pollutants and hospital admissions for chronic obstructive pulmonary disease in Hong Kong. Thorax. 2007 Sep;62(9):780-5. doi: 10.1136/thx.2006.076166. Epub 2007 Feb 20. PMID 17311838
- [Background] Ko FW, Tam W, Tung AH, Ngai J, Ng SS, Lai K, Au KF, Hui DS. A longitudinal study of serial BODE indices in predicting mortality and readmissions for COPD. Respir Med. 2011 Feb;105(2):266-73. doi: 10.1016/j.rmed.2010.06.022. Epub 2010 Jul 22. PMID 20655186
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Halpern MT, Stanford RH, Borker R. The burden of COPD in the U.S.A.: results from the Confronting COPD survey. Respir Med. 2003 Mar;97 Suppl C:S81-9. doi: 10.1016/s0954-6111(03)80028-8. PMID 12647946
- [Background] Seemungal TA, Donaldson GC, Paul EA, Bestall JC, Jeffries DJ, Wedzicha JA. Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1418-22. doi: 10.1164/ajrccm.157.5.9709032. PMID 9603117
- [Background] Donaldson GC, Seemungal T, Jeffries DJ, Wedzicha JA. Effect of temperature on lung function and symptoms in chronic obstructive pulmonary disease. Eur Respir J. 1999 Apr;13(4):844-9. doi: 10.1034/j.1399-3003.1999.13d25.x. PMID 10362051
- [Background] Ko FW, Ng TK, Li TS, Fok JP, Chan MC, Wu AK, Hui DS. Sputum bacteriology in patients with acute exacerbations of COPD in Hong Kong. Respir Med. 2005 Apr;99(4):454-60. doi: 10.1016/j.rmed.2004.09.011. PMID 15763452
- [Background] Manini TM, Everhart JE, Patel KV, Schoeller DA, Colbert LH, Visser M, Tylavsky F, Bauer DC, Goodpaster BH, Harris TB. Daily activity energy expenditure and mortality among older adults. JAMA. 2006 Jul 12;296(2):171-9. doi: 10.1001/jama.296.2.171. PMID 16835422
- [Background] Hamer M, Stamatakis E. Physical activity and mortality in men and women with diagnosed cardiovascular disease. Eur J Cardiovasc Prev Rehabil. 2009 Apr;16(2):156-60. doi: 10.1097/HJR.0b013e32831f1b77. PMID 19276984
- [Background] Waschki B, Kirsten A, Holz O, Muller KC, Meyer T, Watz H, Magnussen H. Physical activity is the strongest predictor of all-cause mortality in patients with COPD: a prospective cohort study. Chest. 2011 Aug;140(2):331-342. doi: 10.1378/chest.10-2521. Epub 2011 Jan 27. PMID 21273294
- [Background] Katz P, Chen H, Omachi TA, Gregorich SE, Julian L, Cisternas M, Balmes J, Blanc PD. The role of physical inactivity in increasing disability among older adults with obstructive airway disease. J Cardiopulm Rehabil Prev. 2011 May-Jun;31(3):193-7. doi: 10.1097/HCR.0b013e3181fc09b7. PMID 21124233
- [Background] van den Borst B, Slot IG, Hellwig VA, Vosse BA, Kelders MC, Barreiro E, Schols AM, Gosker HR. Loss of quadriceps muscle oxidative phenotype and decreased endurance in patients with mild-to-moderate COPD. J Appl Physiol (1985). 2013 May;114(9):1319-28. doi: 10.1152/japplphysiol.00508.2012. Epub 2012 Jul 19. PMID 22815389
- [Derived] Ko FW, Tam W, Siu EHS, Chan KP, Ngai JC, Ng SS, Chan TO, Hui DS. Effect of short-course exercise training on the frequency of exacerbations and physical activity in patients with COPD: A randomized controlled trial. Respirology. 2021 Jan;26(1):72-79. doi: 10.1111/resp.13872. Epub 2020 Jun 15. PMID 32542906